CLINICAL TRIAL: NCT06386016
Title: Detection of Valvular Heart Disease Using Artificial Intelligence-based Stethoscope
Status: Recruiting | Type: Observational
Sponsor: Xiao-dong Zhuang (Other)
Responsible Party: Sponsor-Investigator, Xiao-dong Zhuang, Dr, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: Stethoscope study
Record Dates: First submitted 2024-04-24; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with valvular heart disease
  Interventions: Other: artificial intelligence-based stethoscope
- patients without valvular heart disease
  Interventions: Other: artificial intelligence-based stethoscope

INTERVENTIONS:
Other: artificial intelligence-based stethoscope — artificial intelligence-based stethoscope

SUMMARY:
The aim of this study is to develop a deep learning-based application of heart sounds in the diagnosis of valvular heart disease, which can be used to screen patients with valvular heart disease and promote earlier clinical monitoring and intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age>18 years
2. In the past 1 month, echocardiography was performed to diagnose valvular heart disease (positive group) and echocardiography to exclude valvular heart disease (negative group).
3. Consent to study and be able to sign informed consent

Exclusion Criteria:

1. After prosthetic valve replacement
2. Congenital heart disease (except bilobal aortic valve)
3. Hypertrophic Cardiomyopathy（HCM）
4. Pregnant, lactating women

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with and without valvular heart disease assessed by echocardiography
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
valvular heart disease | 10 months
  Reports therefore graded VHD as none, mild, moderate, severe, or critical, with additional borderline categories (eg, moderate to severe) also allowed

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes